CLINICAL TRIAL: NCT04842877
Title: A Phase II Open-label Study Evaluating Valemetostat Tosylate as a Single Agent in Patients With Relapse/Refractory B-cell Lymphoma
Brief Title: Study of Valemetostat Tosylate as a Single Agent in Patients With Relapse/Refractory B-cell Lymphoma
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The Lymphoma Academic Research Organisation (Other)
Collaborators: Daiichi Sankyo (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VALYM
Record Dates: First submitted 2021-04-07; First posted 2021-04-13 (Actual); Last update posted 2025-01-24 (Actual); Status verified 2025-01

CONDITIONS: Lymphoma, B-Cell
Keywords: relapse; valemetostat tosylate
MeSH Terms: conditions — Lymphoma, B-Cell; Recurrence

STUDY DESIGN:
Intervention Model Description: This is a multicenter, prospective, single arm, non-randomized, open-label, phase 2 clinical study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental arm (Experimental): Experimental arm: Valemetostat tosylate (DS-3201b) is given continuously at 200 mg QD.
  Interventions: Drug: Valemetostat tosylate

INTERVENTIONS:
Drug: Valemetostat tosylate — 200mg QD continuously until disease progression, consent withdrawal, unacceptable drug-related toxicity, lost to follow-up, major protocol deviation, pregnancy, termination by sponsor or death, whichever occurs first.
  Other Names: DS-3201b

SUMMARY:
This is a multicenter, prospective, single arm, non-randomized, open-label, phase 2 clinical study to evaluate safety and efficacy of valemetostat tosylate (DS-3201b) in patients with relapsed or refractory B cell lymphoma with 6 cohorts of patients including 2 biology-driven cohorts. Up to 141 patients will be enrolled in 6 different cohorts (40 patients with aggressive B-cell lymphoma, 41 with follicular lymphoma (FL), 20 with Mantle Cell Lymphoma (MCL) and 20 with other indolent lymphomas, and 20 patients with Hodgkin lymphoma (HL)). FL patients with EZH2 mutant (gain of function mutations) will be enrolled in the cohort 2bis. At least 8 aggressive B-cell lymphoma patients with EZH2 mutant will be enrolled in the cohort 1. The primary endpoint is the overall response rate (ORR) determined by investigator assessment.

DETAILED DESCRIPTION:
Each cycle consists of 28 days. Valemetostat tosylate (DS-3201b) is given continuously at 200 mg once daily (QD). The total duration is expected to be approximately 3 years, assuming an expected enrollment duration of 2 years and a minimum duration of valemetostat tosylate (DS- 3201b) administration of 12 cycles of 28 days for the last enrolled patient.

ELIGIBILITY:
Inclusion Criteria:

1 - Participants with confirmed histological diagnosis of B-cell non-Hodgkin's lymphoma of aggressive B-cell lymphoma (diffuse large B-cell lymphoma-not otherwise specified, primary mediastinal B-cell lymphoma, high grade B-cell lymphoma-not otherwise specified and high grade B-cell lymphoma with MYC and BCL2 and/or BCL6 rearrangement, transformed indolent lymphoma and grade 3b follicular lymphoma), FL (grade 1, 2, 3a), MCL, MZL or other indolent lymphoma (Waldenström macroglobulinemia), or HL according to the World Health Organization (WHO) 2016 classification of hematopoietic and lymphoid tissue.

2. Participant who had progressive disease (PD) or did not have a response (CR or PR) in previous systemic therapy, or relapsed or progressed after previous systemic therapy 3. Participant who has measurable disease by the Lugano criteria (ie longest diameter of a nodal site > 1.5cm and/or longest diameter of an extranodal site > 1.0 cm) 4. Participant who had previous standard therapy with at least: (note: patients having received prior CAR-T therapy can be enrolled):

1. For aggressive B-cell lymphoma : 1 prior line of therapy (in transformed indolent lymphoma patient must have received at least one line of treatment containing an anthracycline-based regimen before of after transformation) containing an anti-CD20 antibody and an anthracycline (unless anthracycline-based therapy is contraindicated) and if patient is considered unable to benefit from intensification treatment with autologous stem cell transplant (ASCT) as defined by at least one of the following criteria:

   * Relapsed following, or refractory to, previous ASCT
   * Ineligible for intensification treatment due to age or significant comorbidity
   * Ineligible for intensification treatment due to failure to mobilize an acceptable number of hematopoietic stem cells
   * Refused intensification treatment and/or ASCT
2. For FL, MZL and other indolent non-Hodgkin's lymphoma (NHL): 2 prior lines of systemic therapy with at least one anti-CD20 monoclonal antibody. Local involved field radiotherapy for limited stage disease is not considered as a previous line. Subjects with prior ASCT may be included. Note: for Splenic Marginal Zone Lymphoma (SMZL), splenectomy is considered as one line; for Extranodal Marginal Zone Lymphoma (ENMZL), Helicobacter pylori eradication is not considered as a previous line.
3. For MCL: 2 prior lines including at least one immunochemotherapy and one BTK inhibitor.
4. For HL: 3 prior lines including at least one line with anthracycline-based chemotherapy (unless anthracycline-based therapy is contraindicated), one line containing brentuximab-vedotin and one line containing an anti-PD1 or anti-PDL1 antibody and must be considered unable to benefit from intensification treatment with autologous stem cell transplant (ASCT) as defined by at least one of the following criteria:

   * Relapsed following, or refractory to, previous ASCT
   * Did not achieve at least a partial response to a standard salvage regimen
   * Ineligible for intensification treatment due to age or significant comorbidity
   * Ineligible for intensification treatment due to failure to mobilize an acceptable number of hematopoietic stem cells
   * Refused intensification treatment and/or ASCT 5. Participant with Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2 6. Adequate renal function defined as calculated creatinine clearance ≥ 40 mL/min per the Cockcroft and Gault formula 7. Adequate bone marrow function:
   * Absolute neutrophil count (ANC) > 1000/mm3 (≥ 1 × 109/L) without growth factor support (G-CSF) for at least 7 days
   * Platelets ≥ 75,000/mm3 (≥ 75 × 109/L) evaluated after at least 7 days since last platelet transfusion
   * Hemoglobin > 8.0 g/dL evaluated after at least 7 days since last transfusion 8. Adequate liver function:
   * Total bilirubin < 1.5 × the upper limit of normal (ULN) except for unconjugated hyperbilirubinemia due to Gilbert's syndrome
   * Alkaline phosphatase (ALP) (in the absence of bone disease), alanine aminotransferase (ALT), and aspartate aminotransferase (AST) < 3 × ULN (< 5 × ULN if subject has liver involvement due to lymphoma) 9. Adequate tissue (surgical excision is recommended) for central pathology review and biological characterisation 10. Patient being successfully tested for EZH2 mutation status at study specific laboratories (for cohort 1, 2 and 2bis) 11. Subjects with a history of hepatitis B or C are eligible on the condition that subjects have adequate liver function and are hepatitis B surface antigen negative and have undetectable serum hepatitis B virus (HBV) DNA and hepatitis C virus (HCV) RNA, respectively.

     12. Females of childbearing potential must agree to use an highly effective birth control methods (defined in §13.6.1) during the following time periods related to this study: 1) for at least 28 days before starting study drug; 2) while participating in the study; 3) dose interruptions; and 4) for at least 3 months after discontinuation of study treatment 13. Males with partners of childbearing potential must agree to use highly effective birth control methods during the study and 3 months after last treatment administration 14. Male and female participant ≥18 years of age at the time of informed consent 15. Patient covered by any social security system (France) 16. Patient who understands and speaks one of the country official language 17. Participant who has provided written consent to participate in the study

Exclusion Criteria:

1. Participant with prior exposure to EZH2 inhibitor
2. Participant with active lymphomatous involvement of the central nervous system (CNS) at screening
3. Any prior treatment-related (ie, chemotherapy, immunotherapy, radiotherapy), clinically significant toxicities have not resolved to ≤ Grade 1 per CTCAE version 5.0, or prior treatment-related toxicities are clinically unstable and clinically significant at time of enrollment.
4. Major surgery within 4 weeks before the first dose of study drug.
5. Inability to take oral medication, or malabsorption syndrome or any other uncontrolled gastrointestinal condition (eg, nausea, diarrhea, or vomiting) that might impair the bioavailability of the drug
6. Subjects currently taking medications that are known moderate or strong CYP3A inducers

   * If currently used, these medications need to be discontinued at least 14 days prior to study drug administration; replacement by alternative medications that are not moderate or strong CYP3A inducers can be considered according to medical need
7. Vaccinated with live, attenuated vaccines within 6 months of enrollment (except COVID vaccine)
8. Use of any standard or experimental anti-cancer drug therapy within 4 weeks or a minimum of 3 half lives of the drug, whatever the shortest prior to first administration of study drug,
9. History of CAR T-cells therapy within 30 days prior to the first dose of study drug
10. History of autologous or allogeneic hematopoietic cell transplantation (HCT) within 90 days prior to the first dose of study drug
11. Patients taking corticosteroids within 2 weeks prior to first administration of study drug, unless administered at a cumulated dose equivalent of prednisone to ≤ 10mg /day (within these 2 weeks).
12. Participant with significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II, uncontrolled arterial hypertension, unstable angina, myocardial infarction, or stroke within 6 months of the first dose of study drug; or cardiac ventricular arrhythmia
13. Subjects with malignancies other than B cell lymphomas except subjects who have been disease-free for 2 years (subjects with a history of a completely resected non-melanoma skin cancer or successfully treated in situ carcinoma are eligible).
14. Positive serology of human immunodeficiency virus (HIV)
15. Participant with prolongation of corrected QT interval using Fridericia's formula (QTcF) to > 470 milliseconds (msec) (obtained on average of 3 ECGs)
16. Participant with venous thrombosis or pulmonary embolism not treated
17. Participant with complications of hepatic cirrhosis, interstitial pneumonia, or pulmonary fibrosis
18. Participant with active infection requiring systemic therapy
19. Woman who are pregnant (positive serum pregnancy test at screening) or breastfeeding
20. Participant who were deemed as inappropriate to participate in the study by the investigator or coinvestigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2021-06-11 (Actual); Primary Completion 2024-12-03 (Actual); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | when mature response rate data have been observed, estimated as no later than 12 months after the last patient in each cohort has received the first dose of study drug
  ORR according to Lugano Response Criteria (2014)

SECONDARY OUTCOMES:
Complete Response Rate (CRR) | After 3 cycles of treatment (each cycle of 28 days, id est (ie) 3 months)
  CRR according to Lugano response Criteria
Complete Response (CR) Rate | After 6 cycles of treatment (each cycle of 28 days, id est (ie) 6 months)
  CRR according to Lugano response Criteria
Complete Response (CR) Rate | After 9 cycles of treatment (each cycle of 28 days, id est (ie) 9 months)
  CRR according to Lugano response Criteria
Complete Response (CR) Rate | After 12 cycles of treatment (each cycle of 28 days, id est (ie) 12 months)
  CRR according to Lugano response Criteria
Progression-Free Survival (PFS) | After 12 cycles(each cycle is 28 days) of study treatment for the last patient included (estimated 3 years of study)
  PFS is defined as the time from inclusion into the study to the first observation of documented clinical disease progression or death due to any cause.
Duration of response (DoR) | After 12 cycles (each cycle is 28 days) of study treatment for the last patient included (estimated 3 years of study)
  The DoR is defined as the time from attainment of CR or PR based on Lugano Response Criteria 2014 to the date of first documented disease progression, relapse (local assessment) or death from any cause
Time to Response (TTR) | After 12 cycles (each cycle is 28 days) of study treatment for the last patient included (estimated 3 years of study)
  The TTR is defined defined as the time from the first dose date to the date of attainment of CR or PR based on Lugano Response Criteria 2014
Number of Serious Adverse Events (SAE) | After 12 cycles of study treatment (each cycle is 28 days) for the last patient included (estimated 3 years of study)
  The frequency of SAE
Pharmacokinetics: quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a) | predose
  quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a)
Pharmacokinetics: quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a) | 1 hour post-dose at Cycle1 Day 1
  quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a)
Pharmacokinetics: quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a) | 2 hours post-dose at Cycle1 Day 1
  quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a)
Pharmacokinetics: quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a) | 4 hours post-dose at Cycle1 Day 1
  quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a)
Pharmacokinetics: quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a) | 5 hours post-dose at Cycle1 Day 1
  quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a)
Pharmacokinetics: quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a) | predose at Cycle1 Day 8
  quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a)
Pharmacokinetics: quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a) | predose at Cycle1 Day 15
  quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a)
Pharmacokinetics: quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a) | predose at Cycle1 Day 22
  quantity of valemetostat tosylate (DS-3201b) and major metabolite (CALZ-1809a)

CONTACTS AND LOCATIONS:
Overall Officials: Franck Morschhauser, PhD, Study Chair — Lymphoma Study Association; Emmanuel Bachy, PhD, Study Chair — Lymphoma Study Association
Locations (22):
- Belgium (4):
  - A.Z. Sint Jan AV, Bruges
  - University Hospital Gent, Ghent
  - CH Tourelle Peltzer, Verviers
  - CHU Mont-Godinne, Yvoir
- France (18):
  - CH d'Avignon, Avignon
  - CH de la Côte Basque, Bayonne
  - Institut Bergonié, Bordeaux
  - Institut d'Hématologie de Basse Normandie, Caen
  - Ch Metropole Savoie - Site Chambery, Chambéry
  - CHU d'Estaing, Clermont-Ferrand
  - François Lemonnier, Créteil
  - CHU de Dijon, Dijon
  - Chd de Vendee, La Roche-sur-Yon
  - Clinique Victor Hugo, Le Mans
  - Service des Maladies du Sang - CHRU de Lille, Lille
  - Institut Paoli Calmette, Marseille
  - CHU de Montpellier, Montpellier
  - Gh Region Mulhouse Et Sud Alsace, Mulhouse
  - CHU Hôtel Dieu, Nantes
  - Emmanuel Bachy, Pierre-Bénite
  - CHU Pontchaillou, Rennes
  - Ch de Bretagne Atlantique -, Vannes

IPD SHARING:
Plan to Share IPD: No